CLINICAL TRIAL: NCT01406535
Title: Sustained Improvement of MYocardial Blood Flow by Intermittent PhosphoDiesterase 5 INhibition in REfractory Coronary ArterY Disease Suggests Enhanced Angiogenesis (SYDNEY)
Brief Title: Improvement of Myocardial Blood Flow by PhosphoDiesterase 5 Inhibition in Coronary Artery Disease
Acronym: SYDNEY
Status: Temporarily not available | Type: Expanded Access
Sponsor: Medical University of Vienna (Other)
Responsible Party: Rudolf Berger, MD, Medical University of Vienna, Department of Internal Medicine, Division of cardiology
Other Study IDs: MUWCard23022011
Record Dates: First submitted 2011-07-29; First posted 2011-08-01 (Estimated); Last update posted 2011-08-01 (Estimated); Status verified 2011-01

CONDITIONS: Therapy Refractory Myocardial Ischemia; Coronary Artery Disease; Unsuitable for Surgical or Percutaneous Revascularisation
Keywords: Phosphodiesterase 5 inhibition; myocardial perfusion; angiogenesis; coronary artery disease; therapy refractory
MeSH Terms: conditions — Coronary Artery Disease | interventions — Vardenafil Dihydrochloride

INTERVENTIONS:
Drug: Vardenafil — 5 mg vardenafil per os twice daily
Other: Placebo — 5 mg placebo per os twice daily

SUMMARY:
The aim of this study is to prospectively investigate if intermittent Phosphodiesterase 5 inhibition for 15 weeks improves myocardial perfusion by angiogenesis in patients with therapy refractory myocardial ischemia due to coronary artery disease judged to be unsuitable for surgical or percutaneous revascularisation. For proof of efficacy the following tests will be performed at baseline and one day and 4 weeks after discontinuation of therapy: Exercise tolerance will be evaluated by bicycle exercise testing. Blood tests will be performed to evaluate markers of angiogenesis (endothelial progenitor cells, vascular endothelial growth factor, basic fibroblast growth factor). The improvement of myocardial perfusion will be tested functionally as increase of coronary flow reserve by positron emission tomography. Moreover, changes in ventricular function, symptoms and quality of life will be assessed.

DETAILED DESCRIPTION:
This study is designed as a randomized, double-blind, placebo controlled monocentric study.

Patients will be randomized to two groups; PDE5 inhibitor (vardenafil) or placebo taken as one tablet twice per day for 15 weeks. The analyses will be performed under blinded conditions by external experts not having any direct contact to the investigators or the patients.

Patients with severe coronary artery disease who are judged to be unsuitable for surgical revascularization because of a bad general state of health or unsuitable for percutaneous revascularization because of the bad morphology of coronary arteries by an expert panel of interventionists and cardiac surgeons are eligible for this study. Eligible patients meeting inclusion criteria will be invited for participation. At the screening visit (Visit -1) demographic data, medical history, and concomitant medication are documented, vital signs are checked, a physical examination, an ECG, and a routine laboratory test is performed. After giving written informed consent for participation in the study, the patient is randomized to one of the two study groups - PDE5 inhibitor (vardenafil) or placebo taken as one pill twice per day for 15 weeks. Within three weeks after this screening visit, baseline efficacy tests are performed. After the last baseline test the study medication is distributed to the patient (Visit 0). During the treatment phase follow-up visits are scheduled after week 1, 3, 6, and 12 (Visit 1-4). Between week 13 and 15 the same efficacy tests as performed at baseline will be repeated. The final visit after the last efficacy test terminates the active study phase at week 15 (Visit 5). During visit 0 to 5 a clinical examination, an ECG, and clinical routine laboratory parameters (blood chemistry, blood cell count, and coagulation parameters) of the patient are performed.

For proof of efficacy the following tests will be performed at baseline and one day and 4 weeks after discontinuation of therapy: Exercise tolerance will be evaluated by bicycle exercise testing. Blood tests will be performed to evaluate markers of angiogenesis (endothelial progenitor cells, vascular endothelial growth factor, basic fibroblast growth factor). The improvement of myocardial perfusion will be tested functionally as increase of coronary flow reserve by positron emission tomography. Moreover, changes in ventricular function, symptoms and quality of life will be assessed.

Endpoints of this study are:

Primary Endpoint:

- Total exercise duration (bicycle exercise testing)

Secondary Endpoints:

* Time to 1mm ST-segment depression (bicycle exercise testing)
* Time to limiting angina (bicycle exercise testing)
* Myocardial blood flow (PET)
* Left ventricular ejection fraction (PET)
* Mean angina frequency per week
* Score Seattle Angina Questionnaire
* Natriuretic peptides

ELIGIBILITY:
Inclusion Criteria:

* Stable angina pectoris
* Evidence for myocardial ischemia according to the presence of one or more of the followings:
* Typical angina during exercise test or
* Significant reversible perfusion defects on dipyridamole myocardial radionuclide study
* Coronary artery disease of at least one large epicardial coronary artery with ≥70% stenosis remaining from which new collaterals/vessels could be supplied
* Coronary artery disease judged to be unsuitable for surgical or percutaneous revascularisation ƒdue to extensive atherosclerosis
* Optimized anti-ischemic drug therapy (including beta-blocker therapy with at least 50% target dose)

Subject must be willing and able to give informed consent Eligible patients must fulfill all 6 inclusion criteria.

Exclusion Criteria:

* STEMI or NSTEMI within the past 3 months
* Revascularisation procedures within the last 3 months
* Severely reduced systolic left ventricular function EF < 30%
* Systolic blood pressure <120mmHg
* Chronic renal insufficiency with a serum creatinine >2.5mg/dl
* Diabetes mellitus with proliferative retinopathy
* Diagnosed or suspected cancer
* Chronic inflammatory disease
* Therapy with nitrates and nicorandil
* Women who are pregnant or lactating
* Patients with a total occluded vessel and reversible perfusion defects at the marginal zone of scare tissue if they have no additional stenosed vessels causing significant reversible perfusion defects.
* Patients with a total occluded vessel and perfusion defect at rest despite evidence of vital myocardium, if they have no additional stenosed vessels causing significant reversible perfusion defects.

Eligible patients must demonstrate none of the exclusion criteria.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Rudolf Berger, MD, Vienna, Vienna, Austria